CLINICAL TRIAL: NCT03243929
Title: Translation of District Sun Safe Policies to Schools
Acronym: SSS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Claremont Graduate University (Other)
Responsible Party: Principal Investigator, Kim D. Reynolds, Principal Investigator, Professor, Claremont Graduate University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 5R01HD074416 (NIH)
Record Dates: First submitted 2017-08-06; First posted 2017-08-09 (Actual); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Sun Safety; Sun Safe Schools; Prevention of Skin Cancer

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): All participants in the Translation of District Sun Safe Policies to Schools arm received 1) initial coaching meeting that guided principals through an evaluation of current sun safety practices, the selection of goals for the implementation of sun safety practices, and guidance on the use of intervention materials to support implementation of sun safety practices in the school, 2) follow-up communications from coaches including email, telephone, and virtual meetings, 3) access to media and online resources to support implementation of sun safety practices, 4) mini-grants to support changes in school sun safety practices.
  Interventions: Behavioral: Translation of District Sun Safe Policies to Schools
- Attention Control (Other): All participants in the attention control arm received three emails during the 20 month intervention period including (1) NASBE's Fit Healthy and Ready to Learn; A School Health Guide Part II: Policies to Promote Sun Safety and Prevent Skin Cancer, (2) CDC's Guidelines for Sun Safety to Prevent Skin Cancer, and (3) a link to the Surgeon General's 2014 Call to Action to Prevent Skin Cancer. This attention-control treatment will equalize schools on awareness of recommendations to implement school sun safety.
  Interventions: Behavioral: Attention Control

INTERVENTIONS:
Behavioral: Translation of District Sun Safe Policies to Schools — Translation of District Sun Safe Policies to Schools intervention was guided by Diffusion of Innovation Theory. Principals and other staff in intervention schools received 1) initial coaching meeting that guided principals through an evaluation of current sun safety practices, the selection of goals for the implementation of sun safety practices, and guidance on the use of intervention materials to support implementation of sun safety practices in the school, 2) follow-up communications from coaches including email, telephone, and virtual meetings, 3) access to media and online resources to support implementation of sun safety practices, 4) mini-grants to support changes in school sun safety practices. These components promoted implementation of the 10 policy components recommended by CDC.
  Arms: Intervention
Behavioral: Attention Control — Schools in the control condition received three emails during the 20 month intervention period including (1) NASBE's Fit Healthy and Ready to Learn; A School Health Guide Part II: Policies to Promote Sun Safety and Prevent Skin Cancer, (2) CDC's Guidelines for Sun Safety to Prevent Skin Cancer, and (3) a link to the Surgeon General's 2014 Call to Action to Prevent Skin Cancer. This attention-control treatment will equalize schools on awareness of recommendations to implement school sun safety.
  Arms: Attention Control

SUMMARY:
The purpose of the Translation of District Sun Safe Policies to Schools study was to test whether schools need assistance to facilitate the implementation of school district board-approved sun safety policies by individual elementary schools. The intervention is expected to produce a change in practices at the school level and to improve the sun safety behavior of children attending the intervention schools compared to control schools. A group of 40 school districts in Southern California that adopted board policy 5141.7 for sun safety provided 118 schools that were randomized to a intervention condition or to an attention control condition. The primary outcome is change in school-level sun safety practices based on 10 Centers for Disease Control and Prevention (CDC) categories for policy change (i.e., sunscreen use, UV protective clothing, hats, student education, teacher education, provision of shade, scheduling to avoid peak UV exposure, parent outreach, resource allocation for sun safety, and an accountability system). This primary outcome was assessed by a survey of the principal and one teacher at each school (N=118 principals and 113 teachers at pretest). Parents (N=1770 at pretest) of children attending the schools completed a self-report measure assessing the secondary outcomes of change in individual-level sun safety behavior of their elementary school aged children and number of communications received from the school regarding sun safety. Assessment of principals, teachers and parents occurred at pretest, just prior to randomization, and at a posttest 20-months after the pretest. One Parent Teacher Association (PTA) representative per school was contacted to assess PTA involvement in intervention activities related to sun safety.

The primary hypothesis was stated for the effectiveness of the intervention condition at increasing school-level sun safety practices consistent with the sun safety policies of the school districts and read, H1: At follow-up, a greater percentage of schools in the intervention condition will implement at least one component of the school district sun safety policy compared to schools randomized to the attention-control condition.

ELIGIBILITY:
Inclusion Criteria:

* School districts in California with school Board Policy 5141.7 available online, and with at least one elementary school.

Exclusion Criteria:

* Schools Districts that do not have school Board Policy 5141.7 online, or do not have any elementary schools

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 118 (Actual)
Dates: Start 2014-01-13 (Actual); Primary Completion 2018-03-21 (Actual); Study Completion 2018-04-10 (Actual)

PRIMARY OUTCOMES:
Measure of implementation of sun safety practices and policy at schools | 20 Months
  Change in implementation of sun safety policy after intervention, through survey administration

SECONDARY OUTCOMES:
Students sun protection behavior | 20 Months
  Change in sun safety behaviors after intervention, through survey administration

CONTACTS AND LOCATIONS:
Overall Officials: Kim D Reynolds, PhD, Principal Investigator — Claremont Graduate University
Locations (1):
- Claremont Graduate University, Claremont, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Reynolds KD, Buller DB, Buller MK, Massie K, Berteletti J, Ashley J, Meenan R. Randomized controlled trial evaluating an intervention supporting implementation of sun safety policies in California public elementary schools. Prev Med. 2020 Aug;137:106125. doi: 10.1016/j.ypmed.2020.106125. Epub 2020 May 7. PMID 32389679